CLINICAL TRIAL: NCT02806557
Title: Profiling Neutrophil Counts in Patients With Cancer During Cycle One of Chemotherapy
Brief Title: Profiling Neutrophil Counts in Patients on Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Dr Geoff Hall, Principal Investigator, University of Leeds
Other Study IDs: MO16/191
Record Dates: First submitted 2016-05-26; First posted 2016-06-20 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Neoplasms; Neutropenia; Febrile Neutropenia
Keywords: Neoplasms; Neutropenia; drug therapy; Hematologic tests; Point-of-care Systems; Febrile neutropenia
MeSH Terms: conditions — Neoplasms; Neutropenia; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- High risk group: Defined as risk of severe neutropenia >20% or risk of neutropenic infective complications >10%, with severe neutropenia defined as absolute neutrophil count <1.0 x10^9/L.
  The intervention is home finger-prick capillary blood count monitoring (up to daily).
  Interventions: Device: Home finger-prick capillary blood count monitoring
- Frequently given regimens: Defined as high number of cases of neutropenia, but risk of severe neutropenia <5%.
  The intervention is home finger-prick capillary blood count monitoring (up to daily).
  Interventions: Device: Home finger-prick capillary blood count monitoring
- Prophylactic GCSF: Patients on primary prophylactic granulocyte colony stimulating factor (GCSF).
  The intervention is home finger-prick capillary blood count monitoring (up to daily).
  Interventions: Device: Home finger-prick capillary blood count monitoring

INTERVENTIONS:
Device: Home finger-prick capillary blood count monitoring — A nurse will visit the participant's home according to the test schedule (up to a maximum frequency of 21 visits in a 21-day cycle) and perform the finger-prick capillary blood test and measure the neutrophil count using the Hemocue® WBC DIFF device.
  Other Names: Hemocue® WBC DIFF

SUMMARY:
The purpose of this trial is to observe the changes in white cell counts in patients with cancer during chemotherapy and to determine if changes in the white cell count in the early days during chemotherapy can be used as a predictor of severe neutropenia and its complications.

DETAILED DESCRIPTION:
Neutropenia is a low count of the type of white blood cells that fight bacterial infection. It is a common toxicity of chemotherapy given for cancer. When complicated by infection, it can necessitate urgent admission to hospital, and can be life-threatening. Recovery of neutrophils is necessary prior to delivery of further chemotherapy. The information available on the changes of neutrophils during chemotherapy is limited by the frequency of blood tests which have historically required a venous blood sample and hence are burdensome to the patient.

There are point-of-care medical devices which measure the white blood cell count from a capillary finger-prick sample, and can be used in the patient's home. The investigators aim to use such a device in this trial to; (i) observe the changes in white cell counts following chemotherapy delivery, (ii) determine if changes in the white cell count in the early days during chemotherapy can be used as a predictor of severe neutropenia and its complications.

This trial forms part of a larger project in which the investigators are exploring the role of home blood count monitoring in the management of severe neutropenia and its complications, and exploring the potential for home blood count monitoring to be used to optimise the dose intensity and density of chemotherapy.

This is a non-randomised trial in adults with solid tumours, recruiting from Leeds Teaching Hospitals NHS Trust only. Consenting participants are required to have regular finger-prick blood tests up to a maximum frequency of daily for the duration of the first cycle of chemotherapy, most commonly 3 weeks. A nurse will visit the participant at home and use the Hemocue® WBC DIFF to perform the test.

This trial is funded by a Technology Strategy Board (Innovate UK) Small Business Research Initiative grant.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumour diagnosis.
* Adults ≥ 18 years.
* Receiving either single agent or combination cytotoxic chemotherapy alone or in combination with other targeted or immunotherapies.
* Participants can be receiving primary prophylactic antibiotics or GCSF.
* Live within boundaries of Local Care Direct service provision.

Exclusion Criteria:

* Inability to give informed consent.
* Concurrent haematological malignancy.
* Known bleeding disorder.
* Known sickle cell disease or β-thalassaemia major.
* Known poorly controlled anti-coagulation (INR >3.5 within 6 months for those on warfarin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with solid tumours receiving systemic anti-cancer therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients from whom sufficient neutrophil counts are obtained during the first cycle of chemotherapy. | 18 months

SECONDARY OUTCOMES:
The proportion of patients who are diagnosed with severe neutropenia (CTCAE v4.0 grade 3 or 4 neutropenia) and its complications. | 18 months
The changes in neutrophil counts early in the first cycle of chemotherapy that determine the risk of severe neutropenia and its complications. | 18 months
  Critical time points for measuring neutrophil counts will be determined dependent upon patterns of neutrophil changes observed and the gradient of neutrophil changes will be categorized according to limits determined by logistic regression modelling and hazard ratio calculations.

OTHER OUTCOMES:
The proportion of patients who decline to enter the study or withdraw from it due to finger-prick capillary sampling. | 18 months
The changes in neutrophil counts early in the first cycle of chemotherapy that determine the risk of severe neutropenia and its complications, when primary prophylactic granulocyte colony stimulating factor is administered. | 18 months
  Critical time points for measuring neutrophil counts will be determined dependent upon patterns of neutrophil changes observed and the gradient of neutrophil changes will be categorized according to limits determined by logistic regression modelling and hazard ratio calculations.
The proportion of patients in whom the neutrophil count does not reach grade 1 neutropenia or worse. | 18 months
The proportion of patients in whom the neutrophil count surpasses the threshold for re-treatment in advance of their planned cycle 2 date. | 18 months
The proportion of patients in whom the neutrophil count is below the threshold for retreatment when cycle 2 is due to be delivered. | 18 months
Estimate cost implications of using home neutrophil count monitoring during chemotherapy using Markov modelling. | 18 months
  The trial data will inform the decision ratios in the Markov model. Aggregated costs associated with each pathway have been calculated using Health Resource grouper software for finished consultant episodes from an audit of patients receiving chemotherapy over a 10 year period at a large Cancer Centre in the United Kingdom. The real numbers and potential numbers in each pathway will be compared to estimate the cost implications.

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Hall, FRCP, PhD, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bodey GP, Buckley M, Sathe YS, Freireich EJ. Quantitative relationships between circulating leukocytes and infection in patients with acute leukemia. Ann Intern Med. 1966 Feb;64(2):328-40. doi: 10.7326/0003-4819-64-2-328. No abstract available. PMID 5216294
- [Background] Rao LV, Ekberg BA, Connor D, Jakubiak F, Vallaro GM, Snyder M. Evaluation of a new point of care automated complete blood count (CBC) analyzer in various clinical settings. Clin Chim Acta. 2008 Mar;389(1-2):120-5. doi: 10.1016/j.cca.2007.12.006. Epub 2007 Dec 14. PMID 18187044
- [Background] Rao, L.V., Moiles, D., Vallero, G.M. and Snyder, M. Finger-Stick Complete Blood Counts: comparison between venous and capillary blood. Point of Care The Journal of Near-Patient Testing & Technology. 2011, 10(3), pp.120-122.
- [Background] Bergh J, Wiklund T, Erikstein B, Lidbrink E, Lindman H, Malmstrom P, Kellokumpu-Lehtinen P, Bengtsson NO, Soderlund G, Anker G, Wist E, Ottosson S, Salminen E, Ljungman P, Holte H, Nilsson J, Blomqvist C, Wilking N. Tailored fluorouracil, epirubicin, and cyclophosphamide compared with marrow-supported high-dose chemotherapy as adjuvant treatment for high-risk breast cancer: a randomised trial. Scandinavian Breast Group 9401 study. Lancet. 2000 Oct 21;356(9239):1384-91. doi: 10.1016/s0140-6736(00)02841-5. PMID 11052580